CLINICAL TRIAL: NCT07226973
Title: A Prospective, Single-Blinded, Partially Randomized Three-Cohort Study Comparing Manual Direct Anterior and Manual Posterior Approaches to a Non-Randomized Robotic Posterior Cohort for Total Hip Arthroplasty Using Gait Analysis
Brief Title: Gait After THA: Direct Anterior vs Manual Posterior vs Robotic Posterior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025.027
Record Dates: First submitted 2025-10-28; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA) of the Hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual Direct Anterior Approach (DAA) (Active Comparator): The DAA utilizes an internervous and intermuscular approach, preserving abductor and posterior soft tissues, and is associated with reduced dislocation rates and accelerated early recovery.⁶ However, it carries a steep learning curve and an elevated risk of lateral femoral cutaneous nerve neuropraxia.
  Interventions: Procedure: Total hip arthroplasty via direct anterior approach (manual, non-robotic)
- Manual Posterior Approach (Active Comparator): PA remains the most commonly used technique worldwide, offering extensile exposure and preserved abductor function, though its historical association with increased dislocation risk has necessitated meticulous capsular and soft-tissue repair.
  Interventions: Procedure: Total hip arthroplasty via posterior approach (manual, non-robotic)
- Robotic-Assisted Posterior Approach (Active Comparator): Robotic-assisted THA introduces computer-navigated precision into implant alignment and biomechanical restoration. Contemporary systems (e.g., MAKO) offer intraoperative haptic guidance and preoperative CT-based planning to improve component placement accuracy.
  Interventions: Procedure: Robotic-assisted total hip arthroplasty via posterior approach

INTERVENTIONS:
Procedure: Total hip arthroplasty via direct anterior approach (manual, non-robotic) — Primary THA performed via a direct anterior approach without robotic assistance
  Arms: Manual Direct Anterior Approach (DAA)
Procedure: Total hip arthroplasty via posterior approach (manual, non-robotic) — Primary THA performed via a posterior approach without robotic assistance
  Arms: Manual Posterior Approach
Procedure: Robotic-assisted total hip arthroplasty via posterior approach — Primary THA via posterior approach using pre-op CT-based planning and intra-op robotic assistance
  Arms: Robotic-Assisted Posterior Approach

SUMMARY:
The purpose of this study is to evaluate the gait biomechanics following THA on 3 groups of subjects undergoing DAA (manual) and PA (manual and robotic) surgical approaches.

DETAILED DESCRIPTION:
Single-center, three-arm, partially randomized interventional study comparing gait biomechanics after primary total hip arthroplasty (THA) via (1) manual direct anterior approach (DAA), (2) manual posterior approach (PA), and (3) robotic-assisted posterior approach (rPA). One surgeon's patients are randomized to DAA vs PA; the second surgeon's patients receive rPA per routine practice. Outcomes assessors are blinded (motion-capture suit conceals dressings/scars). Gait and sit-to-stand analyses are performed pre-op and at 6 and 12 weeks post-op using a Vicon motion capture system with force plates and surface EMG. Patient-reported outcomes are collected with standard instruments. The trial evaluates short-term biomechanical recovery and patient-reported outcomes across approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 undergoing primary elective THA for osteoarthritis
* BMI <35
* Ability to walk unassisted (cane, walker, wheelchair, ect) for > 150 feet preoperatively

Exclusion Criteria:

* Previous hip surgery on the affected side
* Neurological disorders affecting gait
* Contraindication to either DAA or PA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Walking speed during level gait (m/s) | Change from baseline (pre-op) to 6 weeks and 12 weeks post-op.
  Mean self-selected walking speed measured over instrumented walkway during motion-capture trials.
Peak hip abduction moment during stance (Nm/kg) | Change from baseline (pre-op) to 6 weeks and 12 weeks post-op.
  Maximum external hip abduction moment during stance, normalized to body mass.
EMG- Gluteus medius peak activation at initial contact/loading response | Change from baseline (pre-op) to 6 weeks and 12 weeks post-op.
  Peak normalized surface EMG amplitude of the operated-side gluteus medius measured during the initial contact/loading response of level walking. EMG is sampled synchronously with motion capture and force plates, band-pass filtered (~20-450 Hz), rectified, and low-pass filtered (~6 Hz) to form a linear envelope. Strides are time-normalized to 0-100% gait cycle; the peak is extracted within 0-10% of the gait cycle (heel strike through loading response). Amplitude is normalized to the participant's maximum voluntary isometric contraction (%MVIC). Participant-level values are the mean of valid trials at each visit.

SECONDARY OUTCOMES:
postoperative complications-(participants with ≥1 event, %) | through study completion, an average of 1 year
  Postoperative complications include, but are not limited to:
  Surgical & Local Complications Dislocation
  Prosthetic Joint Infection (Early or Late)
  Aseptic Loosening
  Periprosthetic Fracture
  Implant Wear (Osteolysis)
  Wound Complications (Hematoma, Dehiscence)
  Nerve or Vascular Injury
  Leg Length Discrepancy
  Heterotopic Ossification
  Implant Failure or Breakage
  Adverse Local Tissue Reaction (Metallosis)
  Tendon/Muscle Dysfunction
  Medical & Systemic Complications Deep Vein Thrombosis (DVT)
  Pulmonary Embolism (PE)
  Cardiovascular Events (Heart Attack, Stroke)
Patient Reported Outcome Measures-HOOS | Baseline; 6 weeks; 12 weeks; 12 months; change from baseline - Score (0-100)
  Hip Disability and Osteoarthritis Outcome Score. Questionnaire. Range 0-100, higher=better

CONTACTS AND LOCATIONS:
Overall Officials: George Chimento, MD, Principal Investigator — Ochsner Health System
Locations (2):
- United States (2):
  - Ochsner Health Center - Elmwood, Metairie, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varin D, Lamontagne M, Beaule PE. Does the anterior approach for THA provide closer-to-normal lower-limb motion? J Arthroplasty. 2013 Sep;28(8):1401-7. doi: 10.1016/j.arth.2012.11.018. Epub 2013 Mar 16. PMID 23507070
- [Background] Yan L, Ge L, Dong S, Saluja K, Li D, Reddy KS, Wang Q, Yao L, Li JJ, Roza da Costa B, Xing D, Wang B. Evaluation of Comparative Efficacy and Safety of Surgical Approaches for Total Hip Arthroplasty: A Systematic Review and Network Meta-analysis. JAMA Netw Open. 2023 Jan 3;6(1):e2253942. doi: 10.1001/jamanetworkopen.2022.53942. PMID 36719679
- [Background] Higgins BT, Barlow DR, Heagerty NE, Lin TJ. Anterior vs. posterior approach for total hip arthroplasty, a systematic review and meta-analysis. J Arthroplasty. 2015 Mar;30(3):419-34. doi: 10.1016/j.arth.2014.10.020. Epub 2014 Oct 22. PMID 25453632
- [Background] Yoo JI, Cha YH, Kim KJ, Kim HY, Choy WS, Hwang SC. Gait analysis after total hip arthroplasty using direct anterior approach versus anterolateral approach: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2019 Feb 8;20(1):63. doi: 10.1186/s12891-019-2450-2. PMID 30736783
- [Background] Ang JJM, Onggo JR, Stokes CM, Ambikaipalan A. Comparing direct anterior approach versus posterior approach or lateral approach in total hip arthroplasty: a systematic review and meta-analysis. Eur J Orthop Surg Traumatol. 2023 Oct;33(7):2773-2792. doi: 10.1007/s00590-023-03528-8. Epub 2023 Apr 3. PMID 37010580
- [Background] Putananon C, Tuchinda H, Arirachakaran A, Wongsak S, Narinsorasak T, Kongtharvonskul J. Comparison of direct anterior, lateral, posterior and posterior-2 approaches in total hip arthroplasty: network meta-analysis. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):255-267. doi: 10.1007/s00590-017-2046-1. Epub 2017 Sep 27. PMID 28956180
- [Background] Wang Z, Bao HW, Hou JZ. Direct anterior versus lateral approaches for clinical outcomes after total hip arthroplasty: a meta-analysis. J Orthop Surg Res. 2019 Feb 26;14(1):63. doi: 10.1186/s13018-019-1095-z. PMID 30808382
- [Background] Wang Z, Hou JZ, Wu CH, Zhou YJ, Gu XM, Wang HH, Feng W, Cheng YX, Sheng X, Bao HW. A systematic review and meta-analysis of direct anterior approach versus posterior approach in total hip arthroplasty. J Orthop Surg Res. 2018 Sep 6;13(1):229. doi: 10.1186/s13018-018-0929-4. PMID 30189881
- [Background] Fagotti L, Falotico GG, Maranho DA, Ayeni OR, Ejnisman B, Cohen M, Astur DC. POSTERIOR VERSUS ANTERIOR APPROACH TO TOTAL HIP ARTHROPLASTY: A SYSTEMATIC REVIEW AND META-ANALYSIS OF RANDOMIZED CONTROLLED TRIALS. Acta Ortop Bras. 2021 Nov-Dec;29(6):297-303. doi: 10.1590/1413-785220212906244610. PMID 34849093
- [Background] Barrett WP, Turner SE, Leopold JP. Prospective randomized study of direct anterior vs postero-lateral approach for total hip arthroplasty. J Arthroplasty. 2013 Oct;28(9):1634-8. doi: 10.1016/j.arth.2013.01.034. Epub 2013 Mar 19. PMID 23523485
- [Background] Cheng TE, Wallis JA, Taylor NF, Holden CT, Marks P, Smith CL, Armstrong MS, Singh PJ. A Prospective Randomized Clinical Trial in Total Hip Arthroplasty-Comparing Early Results Between the Direct Anterior Approach and the Posterior Approach. J Arthroplasty. 2017 Mar;32(3):883-890. doi: 10.1016/j.arth.2016.08.027. Epub 2016 Aug 31. PMID 27687805
- [Background] Rosenlund S, Broeng L, Holsgaard-Larsen A, Jensen C, Overgaard S. Patient-reported outcome after total hip arthroplasty: comparison between lateral and posterior approach. Acta Orthop. 2017 Jun;88(3):239-247. doi: 10.1080/17453674.2017.1291100. Epub 2017 Feb 18. PMID 28464754
- [Background] Meneghini RM, Smits SA, Swinford RR, Bahamonde RE. A randomized, prospective study of 3 minimally invasive surgical approaches in total hip arthroplasty: comprehensive gait analysis. J Arthroplasty. 2008 Sep;23(6 Suppl 1):68-73. doi: 10.1016/j.arth.2008.05.014. PMID 18722305
- [Background] Petis S, Howard J, Lanting B, Jones I, Birmingham T, Vasarhelyi E. Comparing the anterior, posterior and lateral approach: gait analysis in total hip arthroplasty. Can J Surg. 2018 Feb;61(1):50-57. doi: 10.1503/cjs.003217. Epub 2017 Dec 1. PMID 29368677
- [Background] Reininga IH, Stevens M, Wagenmakers R, Boerboom AL, Groothoff JW, Bulstra SK, Zijlstra W. Comparison of gait in patients following a computer-navigated minimally invasive anterior approach and a conventional posterolateral approach for total hip arthroplasty: a randomized controlled trial. J Orthop Res. 2013 Feb;31(2):288-94. doi: 10.1002/jor.22210. Epub 2012 Aug 8. PMID 22886805
- [Background] Nelms NJ, Birch CE, Halsey DH, Blankstein M, McGinnis RS, Beynnon BD. Assessment of Early Gait Recovery After Anterior Approach Compared to Posterior Approach Total Hip Arthroplasty: A Smartphone Accelerometer-Based Study. J Arthroplasty. 2020 Feb;35(2):465-470. doi: 10.1016/j.arth.2019.09.030. Epub 2019 Sep 26. PMID 31629624